CLINICAL TRIAL: NCT03166241
Title: Serum Interleukin -21 Level in Patients With Severe Adverse Cutaneous Drug Reaction and Correlation With Disease Severity.
Brief Title: Serum Interleukin -21 Level in Patients With Severe Adverse Cutaneous Drug Reaction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAHanna, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACDR
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Adverse Cutaneous Reaction to Alternative Medical Therapy
MeSH Terms: interventions — Liver Function Tests; Blood Sedimentation; Kidney Function Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): measure serum interleukin 21 level in patients with severe adverse drug reaction who show change in serum interleukin 21 before and after therapy the following investigation will be done at the begning of the study to patients: Complete Blood Picture Erythrocyte Sedimentation Rate Random blood sugar Liver function tests Kidney function tests
  Interventions: Diagnostic Test: serum interleukin 21; Diagnostic Test: Complete Blood Picture; Diagnostic Test: Liver function test; Diagnostic Test: Random Blood Sugar; Diagnostic Test: Erythrocyte Sedimentation Rate; Diagnostic Test: Kidney function tests
- control group (Placebo Comparator): compare serum interleukin 21 level in patients with severe adverse drug reaction and healthy control subjects
  Interventions: Diagnostic Test: serum interleukin 21

INTERVENTIONS:
Diagnostic Test: serum interleukin 21 — it is cytokine used as a marker to detect it's level in patients with adverse drug reactions
Diagnostic Test: Complete Blood Picture — It is a blood sample will taken from patients to detect any abnormalities in blood component at the start of the study
  Arms: study group
Diagnostic Test: Liver function test — It is a blood sample will taken from patients to detect any associated liver disease at the start of the study
  Arms: study group
Diagnostic Test: Random Blood Sugar — measure blood sugar in patients included in the study at the start of the study
  Arms: study group
Diagnostic Test: Erythrocyte Sedimentation Rate — blood sample will be taken from patients to detect any abnormalities in erythrocyte sedimentation rate at the start of the study
  Arms: study group
Diagnostic Test: Kidney function tests — blood sample will be taken from patients to detect any kidney disease before the start of the study
  Arms: study group

SUMMARY:
Adverse cutaneous drug reactions are undesirable and typically unanticipated reactions independent of the intended therapeutic purpose of a medication. It may be either immunologic (eg, drug allergy) or non-immunologic. Adverse cutaneous drug reaction produce a wide range of clinical manifestations such as pruritus, maculopapular eruptions, urticaria, angioedema, phototoxic and photo allergic reactions, fixed drug reactions, erythema multiforme,vesiculobullous reactions (eg, Stevens-Johnson syndrome and toxic epidermal necrolysis) and serum sickness .They must be considered in the differential diagnosis of sudden symmetric eruption

DETAILED DESCRIPTION:
Erythema multiforme is an acute immune mediated disorder It is a type IV hypersensitivity reaction leading to dermal vasculitis. Erythema multiforme major usually as a result of medications such as sulphonamides, non-steroidal anti-inflammatories and penicillin and there is skin and mucosal involvement.

Steven-Johnson syndrome (SJS) and Toxic Epidermal Necrolysis (TEN) are considered a spectrum of acute life-threatening mucocutaneous reactions that differ only in severity. Both diseases are characterized by mucous membrane and skin involvement, are often caused by medications and are collectively known as epidermal necrolysis or scalded skin syndrome.Stevens-Johnson syndrome (SJS) is classified as an epidermal loss <10% of the body surface area.Toxic Epidermal Necrolysis (TEN) is indicated by >30% body surface area erosion. The range of epidermal loss between 10% and 30% is called Stevens-Johnson syndrome-Toxic Epidermal Necrolysis (SJS-TEN) overlap. Severity of illness score [Score of Toxic Epidermal Necrolysis(TEN) ] has been devised to predict prognosis in patients with Epidermal Necrolysis.This scoring system addresses 7 prognostic factors: age, malignancy, heart rate,Body Surface Area involved, serum urea, serum glucose and serum bicarbonate levels.

Interleukin-21 regulates both innate and adaptive immune responses and it is not only has key roles in antitumour and antiviral responses that promote the development of autoimmune diseases and inflammatory disorders. It is recently discovered member of the type 1 cytokine family which is produced by activated clusters of differentiation 4+ T cells ,Natural killer cells and follicular helper T cells.

ELIGIBILITY:
Inclusion Criteria:

* 20 patients presenting with adverse cutaneous drug reaction (Erythema multiforme, SJS and TEN )
* Patients with definite drug history.
* Both sex will be included.

Exclusion Criteria:

* Patients with a history of topical or systemic treatment (corticosteroids, intralesional steroid injection, immunosuppressive therapy).
* Patients within 4 weeks of the study.
* Patients receiving phototherapy within 6 months of the study.
* Diabetic patients
* Anaemic patients
* Thyroid disorders,
* Chronic liver or Renal diseases
* Atopy and Parathyroid disorders.
* Patients with known autoimmune diseases or cancer.
* Pregnant or lactating womens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the patients with severe adverse cutaneous drug reaction who show change in serum interleukin 21 before and after therapy | one month
  blood sample will be taken from patients

REFERENCES:
- [Result] Farshchian M, Ansar A, Zamanian A, Rahmatpour-Rokni G, Kimyai-Asadi A, Farshchian M. Drug-induced skin reactions: a 2-year study. Clin Cosmet Investig Dermatol. 2015 Feb 9;8:53-6. doi: 10.2147/CCID.S75849. eCollection 2015. PMID 25709487
- [Result] Hidajat C, Loi D. Drug-mediated rash: erythema multiforme versus Stevens-Johnson syndrome. BMJ Case Rep. 2014 Sep 22;2014:bcr2014205543. doi: 10.1136/bcr-2014-205543. PMID 25246464
- [Result] Ellender RP, Peters CW, Albritton HL, Garcia AJ, Kaye AD. Clinical considerations for epidermal necrolysis. Ochsner J. 2014 Fall;14(3):413-7. PMID 25249808
- [Result] Gong F, Su Q, Pan YH, Huang X, Shen WH. The emerging role of interleukin-21 in allergic diseases (Review). Biomed Rep. 2013 Nov;1(6):837-839. doi: 10.3892/br.2013.166. Epub 2013 Sep 12. PMID 24649038